CLINICAL TRIAL: NCT04690829
Title: Biomarkers in Ocular Inflammation and Uveitis
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000209; 000209-EI
Record Dates: First submitted 2020-12-30; First posted 2020-12-31 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04-15

CONDITIONS: Uveitis; Ocular Inflammation
Keywords: Ocular imaging; Laboratory mARKERS; Natural History
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- control: control with non-inflammatory related eye disease
- control (healthy participant): healthy volunteer
- uveitis: patients with a diagnosis of uveitis or ocular inflammation

SUMMARY:
Background:

Uveitis refers to a large group of inflammatory diseases in the eye. The inflammation can be caused by many factors, such as trauma, medicine, or infection. It can also be caused by systemic diseases. Uveitis and ocular inflammation can cause vision loss. Both children and adults can have uveitis. Standard treatment is to suppress the immune system. But this can result in high costs as well as bad side effects. Researchers want to look at data from NEI studies. They want to learn more about how uveitis progresses and responds to treatment.

Objective:

To find biomarkers to better understand uveitic diseases, assess disease severity, and create outcome measures of response to treatment and disease activity.

Eligibility:

People ages 4 and older from certain NEI studies who have uveitis or ocular inflammation, and healthy volunteers

Design:

Data will be taken from NEI studies from January 1, 2000, to December 31, 2025. Data will only be collected for participants who agreed to let their data be used for future research. No new tests will be done on any samples.

Laboratory results and images will be used. Medical chart data, such as symptoms, medicine history, and treatment course, will be used. Personal data, such as name, medical record number, and date of birth, will be used.

COVID-19 has been reported to cause eye changes. Exam findings of participants who had COVID-19 will be reviewed as well.

Machine learning will be used to study the data.

This study will take place at the NIH Clinical Center. All data will be securely stored.

DETAILED DESCRIPTION:
Study Description: Uveitis refers to a large group of intraocular inflammatory diseases that can cause devastating visual loss in adults and children. This is a retrospective study to identify factors and biomarkers that are relevant to the pathogenesis, progression, and treatment response in inflammatory eye conditions.

Objectives:

The primary objective is to identify ocular imaging, clinical and laboratory biomarkers in order to better classify presentations of uveitic diseases, assess disease severity and develop outcome measures of response to treatment. The secondary objectives are to identify etiological factors for uveitic diseases including through using a machine-learning approach with external collaborators.

Study Population: The study population will be any patient with a diagnosis of uveitis or ocular inflammation enrolled in an IRB approved protocol since 2000.

Description of Sites/Facilities conducting research: Research will be conducted at the National Institutes of Health clinical center

Study Duration: Estimated study duration is 5 years

ELIGIBILITY:
* INCLUSION CRITERIA:

The study population will include subjects aged 4 or older and no upper limit for age will be set. All data will be derived only from subjects evaluated at the NEI eye clinic and enrolled in NEI protocols. This also applies to data from healthy volunteers.

1. Subjects evaluated under the IRB protocols.

   AND
2. Have a diagnosis of uveitis, ocular inflammation, scleritis or a disease known to be associated with intraocular inflammation, (e.g., sarcoidosis, Beh(SqrRoot)(Beta)et s disease, multiple sclerosis (MS) and lymphoma or COVID-19 or other infections)

   OR
3. Serve as a control:

   1. unaffected control (healthy volunteer) or
   2. control with non-inflammatory related eye disease

EXCLUSION CRITERIA:

1. Patients without appropriate diagnostic and laboratory investigations for their diagnosis. Disease specific exclusion criteria will also be used. Patients will be excluded if appropriate laboratory investigations were not performed such as infectious serological tests and autoimmune labs. For posterior segment uveitis with retinal vasculitis, patients without fluorescein angiography will be excluded. Similarly, patients with choroiditis will be excluded if fundus autofluorescence studies were not performed. These disease specific exclusion criteria do not apply to healthy volunteers.

Patients who were minors and NIH employees will be included in this retrospective study. The IRB approved protocols which these patients were managed under allow for the inclusion of these populations at time of original consent.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants evaluated at the NIH clinical center under a NIH approved protocol
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
identify associations in laboratory markers | at baseline
  identify associations in laboratory markers with disease etiology
changes in ocular imaging findings | pre- and post treatment
  changes in ocular imaging findings including as OCT, OCTA, FA, ICG

CONTACTS AND LOCATIONS:
Overall Officials: Tiarnan DL Keenan, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States